CLINICAL TRIAL: NCT00003951
Title: A Phase II Study of Intravenous DX-8951f Administered Daily for Five Days Every Three Weeks to Patients With Metastatic Carcinoma of the Pancreas
Brief Title: DX-8951f in Treating Patients With Metastatic Cancer of the Pancreas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000067147; DAIICHI-8951A-PRT009; JHOC-99062405; MSKCC-99014
Record Dates: First submitted 1999-11-01; First posted 2004-08-18 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Pancreatic Cancer
Keywords: recurrent pancreatic cancer; duct cell adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — exatecan

INTERVENTIONS:
Drug: exatecan mesylate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of DX-8951f in treating patients who have metastatic cancer of the pancreas that has not been previously treated or that has not responded to previous chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the objective response rate in patients with metastatic carcinoma of the exocrine pancreas treated with DX-8951f. II. Determine the time to tumor progression in patients receiving this drug. III. Determine the survival at 6 and 12 months of patients receiving this drug. IV. Evaluate the quantitative and qualitative toxicities of this regimen in this patient population. V. Evaluate the pharmacokinetics of this drug in this patient population.

OUTLINE: Patients receive DX-8951f IV over 30 minutes daily for 5 days. Courses repeat every 21 days. Treatment continues in the absence of unacceptable toxicity or disease progression. Patients are followed every 3 months until death.

PROJECTED ACCRUAL: A total of 12-37 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed epithelial cancer of the exocrine pancreas Metastatic disease Previously untreated disease or progressive disease after first-line chemotherapy Bidimensionally measurable disease Indicator lesion must be outside of any prior radiation port No brain metastases No islet cell tumors, lymphoma, or sarcoma of the pancreas

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT/SGPT no greater than 2 times upper limit of normal (ULN) (5 times ULN if liver metastases present) Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: No active congestive heart failure No uncontrolled angina No myocardial infarction within the past 6 months Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No concurrent serious infection No history of other malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix No overt psychosis, mental disability, or incompetence No other life threatening illness

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent biologic therapy No prophylactic colony stimulating factors to prevent neutropenia Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy and recovered No other concurrent cytotoxic chemotherapy Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiotherapy and recovered No concurrent radiotherapy Surgery: At least 4 weeks since prior major surgery and recovered No concurrent surgery Other: No other concurrent anticancer treatment At least 28 days since other prior investigational drugs, including analgesics or antiemetics No other investigational drugs during and for 28 days after study No concurrent drugs that induce or inhibit CYP3A enzyme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 1999-06; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L. DeJager, MD, FACP, Study Chair — Daiichi Sankyo
Locations (3):
- United States (3):
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas